CLINICAL TRIAL: NCT01810445
Title: Endoscopic Subsurface Optical Imaging for Cancer Detection
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 200210092-9; Endoscopic Subsurface Study
Record Dates: First submitted 2011-08-02; First posted 2013-03-13 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; Laser; Optical
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Patients undergoing a surgical bladder procedure in the main O.R.

SUMMARY:
The purpose of this pilot study is to develop the methodology for an innovative subsurface imaging technology that was designed at Lawrence Livermore National Laboratory. It will allow the non-invasive analysis and imaging of tissues and chemical distributions in the body at an imaging depth of up to 1 centimeter with spatial resolution on the order of 1 mm.

DETAILED DESCRIPTION:
This is a pilot, feasibility study to determine if the subsurface imaging technology warrants advancement to a larger clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be scheduled for a bladder procedure (TURBT or Cystectomy) at the University of California Davis Medical Center.

Exclusion Criteria:

* Non bladder surgical procedures at University of California Davis Medical Center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients already scheduled to undergo a bladder surgery at UCDMC.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 1999-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Accuracy of the subsurface laser to determine cancer cells versus normal cells when viewed endoscopically during a surgical procedure. | 1 year
  Does the subsurface laser allow enough light to visually assess the cells. Logical metric of either "Yes" or "No".

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Demos, PhD, Principal Investigator — University of California, Davis